CLINICAL TRIAL: NCT04313842
Title: A Clinical Study to Explore the Feasibility of AVATAMED in Predicting the Cilnical Response to Temozolomide in Glioblastoma Patients, a Single-center, Prospective Study
Brief Title: A Explorative Study to Evaluate the Clinical Feasibility of AVATAMED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Doo-Sik Kong (Other)
Responsible Party: Sponsor-Investigator, Doo-Sik Kong, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Other Study IDs: 2018-12-071
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: AVATAMED — tumor specimen will be sent for in vitro drug screening experiment and the result will be analyzed by 'AVATAMED' to predict the clinical response

SUMMARY:
This is an exploratory study to evaluate the clinical feasibility of medical deivce 'AVATAMED' for predicting the clinical response to TMZ (temozolomide) in glioblasotma patients.

DETAILED DESCRIPTION:
Glioblastoma patients who would take TMZ treatment will be screened for in vitro drug screening experiment. Patients whose tumor specimen pass the drug screening process will be finally enrolled.

Actual clinical response to TMZ treatment will be compared to drug screening results derived from AVATAMED, a medical software device to predict the drug response based on in vitro assay using patient-derived tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent
2. histologically confirmed glioblastoma patients who will take TMZ treatment
3. KPS >70
4. adequte end-organ function
5. prior major surgery > 4 weeks (prior minor surgery > 1weeks)
6. prior standard concurrent chemo-radiation therapy > 4 weeks
7. prior radiation therapy (including stereotactic radiosurgery) > 12 weeks

Exclusion Criteria:

1. contraindication to TMZ
2. prior anti-cancer therapy except standard of care (*standard of care includes surgery, Stupp regimen, and radiotherapy)
3. uncontrolled systemic medical illness
4. pregnancy

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: among histologically confirmed glioblastoma patients, patients with samples which passed the QC screening process of in vitro drug screening experiment will be finally enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
6 month PFS rate | 6 month
  the fraction of patients without disease progression at 6 months after the TMZ treatment

CONTACTS AND LOCATIONS:
Overall Officials: Doo-sik Kong, MD PhD, Principal Investigator — Professor
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided